CLINICAL TRIAL: NCT02043691
Title: Evaluation of All-Cause Mortality and Pulmonary Morbidity in Treating Juxtarenal, Suprarenal, Thoracoabdominal, and Aortic Arch Pathologies Using Cook Custom Aortic Endografts, the Zenith t-Branch Endovascular Graft, and the Surgeon-Modified Endograft
Brief Title: Evaluation of the Cook Custom Aortic Endograft, the Zenith t-Branch Endovascular Graft, and Surgeon-Modified Endograft in Treating Aortic Pathologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Principal Investigator, Adam W Beck, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201400001
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Juxtarenal Aortic Aneurysm; Suprarenal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm; Penetrating Aortic Ulcer; Aortic Arch Aneurysm; Aortic Dissection
Keywords: Endovascular; Aortic; Aneurysm; Thoracoabdominal; Juxtarenal; Suprarenal; Endograft; Fenestrated; Branched; Complex; Abdominal; Thoracic; Stent; Stentgraft; Arch; Ascending; Dissection; Descending
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Penetrating Atherosclerotic Ulcer; Aneurysm, Aortic Arch; Aortic Dissection; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cook Custom Aortic Endograft (Experimental): Participants will receive the following: (Juxtarenal, Suprarenal, Thoracoabdominal) Clinical Exam, Blood Tests, CT Scans (with and without contrast) or Ultrasound, Abdominal Device X-ray, and Angiography. (Aortic Arch) Clinical Exam, Neurological Exam, Blood Tests, Echocardiogram, CT Scans (with and without contrast), Chest X-ray, and Angiography.
  These tests will aid in the design of the Cook Custom Aortic Endograft. The Cook Custom Aortic Endograft has a variable design such that seal and fixation may be obtained proximal and distal to pathology in the juxtarenal aorta, suprarenal aorta, thoracoabdominal aorta, or the aortic arch aorta. Grafts may include a combination of up to 5 fenestrations and/or branches.
  Interventions: Device: Cook Custom Aortic Endograft
- Zenith t-Branch Endovascular Graft (Experimental): Participants will receive the following: Clinical Exam, Blood Tests, CT Scans (with and without contrast) or Ultrasound, Abdominal Device X-ray, and Angiography. These tests will aid in the sizing of the the Zenith t-Branch Endovascular Graft. The Zenith t-Branch Endovascular Graft is a tubular graft with four branches and a covered stent at the proximal end that contains barbs for proximal fixation of the device. The graft is designed to be connected with celiac, superior mesenteric and two renal arteries via self-expanding covered bridging stents.
  Interventions: Device: Zenith t-Branch Endovascular Graft
- Surgeon-Modified Endograft (Experimental): Participants will receive the following: Clinical Exam, Blood Tests, CT Scans (with and without contrast) or Ultrasound, Abdominal Device X-ray, and Angiography. These tests will aid in the design of the Surgeon-Modified Endografts. These will be created in the operating room by modifying a commercially-available Cook Alpha Thoracic Endograft or Cook Zenith Infrarenal Aortic Device such that seal and fixation may be obtained proximal and distal to pathology in the juxtarenal aorta, suprarenal or thoracoabdominal aorta. Grafts may include a combination of up to 5 fenestrations and branches.
  Interventions: Device: Surgeon-Modified Endograft

INTERVENTIONS:
Device: Cook Custom Aortic Endograft — The Cook Custom Aortic Endograft has a variable design such that seal and fixation may be obtained proximal and distal to pathology in the juxtarenal aorta, suprarenal aorta, thoracoabdominal aorta, or the aortic arch aorta. Grafts may include a combination of up to 5 fenestrations and/or branches.
  Arms: Cook Custom Aortic Endograft
Device: Zenith t-Branch Endovascular Graft — The Zenith t-Branch Endovascular Graft is a tubular graft with four branches and a covered stent at the proximal end that contains barbs for proximal fixation of the device. The graft is designed to be connected with celiac, superior mesenteric and two renal arteries via self-expanding covered bridging stents.
  Arms: Zenith t-Branch Endovascular Graft
Device: Surgeon-Modified Endograft — The Surgeon-Modified Endografts are created in the operating room by modifying a commercially-available Cook Alpha Thoracic Endograft or Cook Zenith Infrarenal Aortic Device such that seal and fixation may be obtained proximal and distal to pathology in the juxtarenal aorta, suprarenal or thoracoabdominal aorta. Grafts may include a combination of up to 5 fenestrations and branches.
  Arms: Surgeon-Modified Endograft

SUMMARY:
This is a single-center study to evaluate the safety and effectiveness of three investigational devices, the Cook Custom Aortic Endograft, the Zenith t-Branch Endovascular Graft, and the Surgeon-Modified Endografts in the treatment of Juxtarenal, Suprarenal, Thoracoabdominal, and Aortic Arch pathologies involving the at least one brachiocephalic artery or visceral vessels.

The three investigational devices offer an endovascular approach to treat complex aortic pathologies that cannot be treated with commercially available devices. This customized, endovascular approach has the potential to decrease hospital length of stay, pulmonary complications, and in-hospital mortality.

DETAILED DESCRIPTION:
Described as follows: Juxtarenal, Suprarenal, Thoracoabdominal aortic pathologies involving at least one visceral artery. Aortic Arch pathologies involving the at least one brachiocephalic artery.

Once the participant has signed the approved informed consent the following tests will be done to determine final subject eligibility and which device will be used:

Juxtarenal, Suprarenal, Thoracoabdominal: Clinical Exam, Blood Tests, CT Scans (with and without contrast), Abdominal Device X-ray, and Angiography.

Aortic Arch: Clinical Exam, Neurological Exam, Blood Tests, Echocardiogram, CT Scans (with and without contrast), Chest X-ray, and Angiography.

The participants will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Juxtarenal, suprarenal, and thoracoabdominal aortic pathology as follows in hemodynamically stable patients:

  1. Intact or contained ruptured aortic or aortoiliac aneurysms (atherosclerotic/degenerative or saccular) involving or in close approximation to the visceral segment of the aorta.

     1. Diameter > 5.5 cm if asymptomatic, or 5.0 cm with enlargement of > 0.5 cm in 6 months.
     2. History of growth > 0.5 cm per year
     3. Any size if ruptured or symptomatic
  2. Penetrating aortic ulcer (PAU)

     1. > 2.0 cm in depth
     2. Any size if contained ruptured or symptomatic
  3. Subacute (>14 days) or chronic (>20 days) aortic dissection with aneurysmal degeneration with at least one of the following:

     1. Total aortic diameter > 5.5 cm if asymptomatic
     2. Total aortic diameter > 4.5 cm if symptomatic
     3. Total aortic diameter > 5.0 cm and history of growth > 0.5 cm in 6 months
* Aortic Arch pathology:

  1. Aneurysm, Ascending thoracic aortic pseudoaneurysm, Type A thoracic aortic dissection, Retrograde type A thoracic aortic dissection between the Sinus of Valsalva and the innominate artery orifice (without involvement of the Aortic Valve), or Ascending penetrating aortic ulcer with and without intramural hematoma
  2. Suitable iliac artery and brachial artery access
  3. Absence of severe landing zone (> 90 degree) angulation that would preclude necessary device delivery/seal/fixation.
  4. Suitable iliac artery access to accommodate device delivery system.
  5. Target arteries for arch branches:

     1. < 24 mm diameter
     2. Adequate landing zone length to obtain proximal and distal seal.
     3. Free from dissection precluding adequate seal in distal landing zone of branch stent and severe tortuosity/thrombus/calcification.
* Aortic Arch Aneurysm

  1. Proximal aortic fixation zone:

     1. Native aorta or surgical graft
     2. Diameter: 20 - 42 mm
  2. Proximal neck length > 20 mm
  3. Must occur distal to coronary arteries and any coronary artery bypass grafts that are considered patent and necessary for proper cardiac perfusion.
  4. Distal aortic fixation zone:

     1. Native aorta or surgical graft
     2. Diameter: 20 - 44 mm
  5. Distal neck length > 20 mm. However, if dissection, distal graft may land in dissected aorta.
  6. Supra-aortic trunk (brachiocephalic) vessels (Any combination of arteries may be used for repair) A. Innominate artery

     1. Native vessel or surgical graft
     2. Diameter: 8 - 22 mm
     3. Length of sealing zone > 10 mm
     4. Acceptable tortuosity B. Left (or right) common carotid artery

     <!-- -->

     1. Native vessel or surgical graft
     2. Diameter 5 - 20 mm
     3. Length of sealing zone > 10 mm C. Left (or right) subclavian artery

     <!-- -->

     1. Native vessel or surgical graft
     2. Diameter 5 - 20 mm
     3. Length of sealing zone > 10 mm
* Aortic Dissection

  1. Access into the true lumen from the groin and at least one supra-aortic trunk vessel.
  2. Seal zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stent-graft would be anticipated to seal off the dissection lumen.
  3. Seal zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen or surgically created.
  4. True lumen size large enough to deploy the device and still gain access into the target branch.

General Exclusion Criteria:

* Less than 18 years of age
* Life expectancy less than 12 months based on the surgeon's assessment
* Pregnant or breastfeeding or planning on becoming pregnant within 60 months
* Inability or refusal to give informed consent
* Unwilling or unable to comply with the follow-up schedule
* Less than 30 days beyond primary endpoint for other investigative drug or device study

Medical Exclusion Criteria:

* Known allergy to the device components (i.e. stainless steel, polyester, solder, gold, or nitinol)
* History of anaphylactic reaction to contrast material that cannot be adequately premedicated
* Systemic or local infection that may increase the risk of endovascular graft infection.
* Baseline eGFR < 30 mL/min (calculated by the Modification of Diet in Renal Disease formula) and not on hemo- or peritoneal dialysis. If the patient is currently on dialysis, or is currently planning on initiating dialysis, then they may undergo repair.
* Body habitus that would inhibit X-ray visualization of the aorta.
* Major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤ 30 days of the endovascular repair.
* Unstable angina, defined as a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina.
* Irreversible coagulopathy

Anatomical Exclusion Criteria:

* Aortic transection due to acute trauma.
* Infectious ("mycotic") etiology of the aortic disease.
* Significant occlusive disease or tortuosity precluding delivery of the device components.
* Juxtarenal, Suprarenal, and Thoracoabdominal:
* Proximal Landing zone < 20 mm in length. The proximal landing zone can be within zones 2 through 8, with least 20 mm of proximal seal and fixation in aorta or Dacron.
* Proximal neck, defined as the thoracic aorta distal to the native left carotid artery, measured outer wall to outer wall on a sectional image (CT) > 41 mm in diameter or < 18 mm in diameter
* Distal landing zone < 20 mm in length if the landing zone is in the aorta, or < 20 mm if the landing zone is in the iliac arteries or in Dacron (in the event the patient has had a previous or concomitant aortic or aorto-iliac reconstruction).
* Untreatable branch vessel stenosis.
* Anatomy that would not allow maintenance of at least one patent hypogastric artery.
* Signs that the inferior mesenteric artery (IMA) is indispensable (i.e. angiographic visualization or a large IMA, filling of superior mesenteric artery (SMA) via collaterals, stenosis of celiac or SMA or oblique views) and the indispensable IMA is not amenable to treatment with a graft branch or fenestration.
* Branching, duplication, aneurysm or untreatable stenosis of the celiac, SMA or renal arteries that would preclude implantation of the investigational devices.
* Aortic arch:
* Proximal neck > 44 mm or < 28 mm in diameter
* Inadequate landing zone to allow adequate distal seal of exclusion of false lumen perfusion in dissection.
* Untreatable branch vessel stenosis.
* Significant occlusive disease, tortuosity, or calcification that would prevent endovascular access.
* Patients qualifying for an industry-sponsored study allowing for a similar repair will be enrolled in the industry-sponsored study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse events at 30 days post primary procedure | 30 days post primary procedure

SECONDARY OUTCOMES:
Rate of all-cause mortality in peri-operative period | Peri-operative
Rate of all-cause mortality at 30 days post primary procedure | 30 days post primary procedure
Number of major adverse events at 6 months post primary procedure | 6 months post primary procedure
Number of subjects requiring ventilation more than 48 hours in peri-operative period | Peri-operative
Average length of ventilation past 48 hours in peri-operative period | Peri-operative
Number of subjects requiring reintubation in peri-operative period | Peri-operative
Average ICU length of stay in peri-operative period | Peri-operative
Number of patients who underwent tracheostomy to treat pulmonary failure at 30 days post primary procedure | 30 days post primary procedure
Number of patients who developed postoperative pneumonia at 30 days post primary procedure | 30 days post primary procedure
Number of patent treated branch vessels at 30 days post primary procedure | 30 days post primary procedure
Number of patients with loss of device integrity at 30 days post primary procedure | 30 days post primary procedure
Freedom from reintervention at 30 days post primary procedure | 30 days post primary procedure
Number of subjects that achieve treatment success at 12 months post procedure | 12 months post procedure
  Treatment success is defined as procedural technical success and patent treated branch vessels at 12 months post procedure, device integrity, and freedom from both reintervention and aortic enlargement ≤5mm as compared to baseline at 12 months post primary procedure.
  Technical success is defined as successful exclusion of the diseased aortic segment without a clinically significant type I or type III endoleak and patent treated branch vessels at the end of the procedure without the need for unanticipated corrective interventions.
Number of major adverse events at 12 months post procedure | 12 months post primary procedure
Number of major adverse events at 2 years post primary procedure | 2 years post primary procedure
Number of major adverse events at 3 years post primary procedure | 3 years post primary procedure
Number of major adverse events at 4 years post primary procedure | 4 years post primary procedure
Number of major adverse events at 5 years post primary procedure | 5 years post primary procedure
Number of patients who underwent tracheostomy to treat pulmonary failure at 6 months post primary procedure | 6 months post primary procedure
Number of patients who underwent tracheostomy to treat pulmonary failure at 12 months post primary procedure | 12 months post primary procedure
Number of patients who developed postoperative pneumonia at 6 months post primary procedure | 6 months post primary procedure
Number of patients who developed postoperative pneumonia at 12 months post primary procedure | 12 months post primary procedure
Number of patent treated branch vessels at 6 months post primary procedure | 6 months post primary procedure
Number of patent treated branch vessels at 12 months post primary procedure | 12 months post primary procedure
Number of patent treated branch vessels at 2 years post primary procedure | 2 years post primary procedure
Number of patent treated branch vessels at 3 years post primary procedure | 3 years post primary procedure
Number of patent treated branch vessels at 4 years post primary procedure | 4 years post primary procedure
Number of patent treated branch vessels at 5 years post primary procedure | 5 years post primary procedure
Number of patients with loss of device integrity at 6 months post primary procedure | 6 months post primary procedure
Number of patients with loss of device integrity at 12 months post primary procedure | 12 months post primary procedure
Number of patients with loss of device integrity at 2 years post primary procedure | 2 years post primary procedure
Number of patients with loss of device integrity at 3 years post primary procedure | 3 years post primary procedure
Number of patients with loss of device integrity at 4 years post procedure | 4 years post procedure
Number of patients with loss of device integrity at 5 years post primary procedure | 5 years post primary procedure
Freedom from reintervention at 6 months post primary procedure | 6 months post primary procedure
Freedom from reintervention at 12 months post primary procedure | 12 months post primary procedure
Freedom from reintervention at 2 years post primary procedure | 2 years post primary procedure
Freedom from reintervention at 3 years post primary procedure | 3 years post primary procedure
Freedom from reintervention at 4 years post primary procedure | 4 years post primary procedure
Freedom from reintervention at 5 years post primary procedure | 5 years post primary procedure
Number of major adverse events at 30 days post primary procedure | 30 days post primary procedure
Rate of neurologic morbidity in peri-operative period | Peri-operative
Rate of neurologic morbidity at hospital discharge | Peri-operative
Rate of neurologic morbidity at 30 days post primary procedure | 30 days post primary procedure
Rate of neurologic morbidity at 6 months post primary procedure | 6 months post primary procedure
Rate of neurologic morbidity at 12 months post primary procedure | 12 months post primary procedure
Rate of neurologic morbidity at 1 year post primary procedure | 1 year post primary procedure
Rate of neurologic morbidity at 2 year post primary procedure | 2 year post primary procedure
Rate of neurologic morbidity at 3 year post primary procedure | 3 year post primary procedure
Rate of neurologic morbidity at 4 year post primary procedure | 4 year post primary procedure
Rate of neurologic morbidity at 5 year post primary procedure | 5 year post primary procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Beck, MD, Principal Investigator — University of Alabama at Bimingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239